CLINICAL TRIAL: NCT04584346
Title: Acute Effects of Medium Chain Triglyceride (MCT) Nutritional Ketosis on Parkinson s Disease (PD) Symptoms and Biomarkers (MCT-PD)
Brief Title: Acute Effects of Medium Chain Triglyceride (MCT) Nutritional Ketosis on Parkinson's Disease (PD) Symptoms and Biomarkers (MCT-PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200153; 20-N-0153
Record Dates: First submitted 2020-10-10; First posted 2020-10-14 (Actual); Results first posted 2022-08-12 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2021-10-13

CONDITIONS: Parkinson's Disease
Keywords: MCT Medium Chain Triglyceride; Ketogenic Diet; Nutritional Ketosis; Parkinson's Biomarkers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Ketogenic Diet
  Interventions: Dietary Supplement: Liquigen MCT oil
- Arm B (Active Comparator): Standard American Diet
  Interventions: Other: Standard American Diet

INTERVENTIONS:
Dietary Supplement: Liquigen MCT oil — MCT oil is a nutritional supplement. The Ketogenic diet restricted carbohydrates to reach 80/5-10/10-15 (lipid:carb:protein daily energy) values
  Arms: Arm A
Other: Standard American Diet — Standard diet with macronutrient composition lipid 35%, protein 10-15%, carbohydrate 50-55%
  Arms: Arm B

SUMMARY:
Background:

The ketogenic diet uses fats as a person's major energy source rather than carbohydrates. There is increasing interest in using this diet to treat neurodegenerative disorders like Parkinson's disease. Researchers want to learn more about the ketogenic diet before recommending this diet in clinical practice.

Objective:

To study the effects of a ketogenic diet for someone with PD.

Eligibility:

People over age 50 with mild to moderate PD.

Design:

Participants will be screened with surveys and a 10-foot walking test. They will have a medical history, physical exam, and blood test.

Participants will be contacted twice in a 1-week period to discuss what they ate over the last 24 hours. They will log data about their daily exercise and activities using an online fitness tracking app.

Participants will stay at NIH Clinical Center for 1 week. They will be put into 1 of 2 groups. One group will follow a ketogenic diet and take MCT oil. The other group will follow a low-fat diet. Their body measurements will be taken. They will meet with a physical therapist and nutritionist.

Participants will have daily respiratory and glucose monitoring. They will have cognitive tests and complete surveys. They will have walking, motor function, and reaction time/finger tapping tests. They will have heart and nerve function tests. They will have electrocardiograms and electroencephalograms. Blood will be taken twice daily.

Participants will follow the ketogenic diet at home for 2 weeks. They will log their activities using the fitness tracking app. Then they will have a follow-up visit at NIH.

Participation in the trial will last for 4 weeks.

DETAILED DESCRIPTION:
Study Description:

While three pilot studies of ketogenic diet (KD) in PD have shown either reduction in motor scores (UPDRS) or improved cognition (memory/fluency), there are gaps in knowledge of the time course and mechanisms of reported outcomes. Furthermore, only a standard ketogenic diet was studied while there are variations such as MCT oil supplementation shown to increase keto-induction, and other adaptations may improve tolerability and micronutrient content. It is the goal of this proposed inpatient metabolic study to address the initial question of effect size and time course of ketosis. If suggestive of benefit in PD, this pilot study may lead to a subsequent larger study of long-term feasibility and effects on disease biomarkers and disease progression, which might also compare alternate diets of interest in PD such as Mediterranean diet. Thus, a pilot feasibility study is proposed, targeting retention rate >80% and adherence in the outpatient setting. Recruitment of 32 participants is based upon power analysis of secondary outcome, testing the Timed Up & Go mobility test that has reported validity in fall prediction, additionally plotting continuous and serially repeated direct/indirect ketosis measurements and motor as well as non-motor symptoms / exploratory disease biomarkers. It is hypothesized that, compared to a non-ketogenic, standard American diet (SAD, also referred to interchangeably as usual diet, ketogenic diet supplemented by MCT oil (MCT-KD) will improve mobility tested by Timed Up & Go (TUG), as well as akinesia, tremor, and memory/executive function tasks, and will reduce motor and non-motor fluctuations within the acute period of keto-induction and early ketogenic timepoints due to improved mitochondrial function and neurotransmitter signaling.

Objectives:

The primary objective is to test the hypothesis that nutritional ketosis (NK) supplemented by MCT oil in a PD cohort (MCT-KD) is feasible for a duration of three weeks. The secondary objective is to show that NK improves PD symptomatology in cognition (improved attention, recall, and executive function), mobility (TUG), and motor function (bradykinesia, akinesia and tremor) within three weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Must be able to speak English
2. Able and willing to provide informed consent
3. Male or female older than age 50 years
4. Clinically probable diagnosis of Parkinson s Disease by UK Brain Bank Criteria, of moderate severity, with ability to safely walk independently for at least a short distance (20 feet) as determined on screening visit
5. BMI > 18.5, to minimize potential risk from expected mild weight loss from ketogenic diet
6. eGFR > 60 by MDRD equation (established on screening visit serum chemistry)
7. MOCA > 20, as well as having in the investigators' assessment the ability and willingness to adhere to either of the study diets
8. Agreement to adhere to Lifestyle Considerations throughout study duration
9. Adhering to Usual Diet (SAD) at baseline, as per investigator determination

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Atypical Parkinsonism or symptoms suggestive of a diagnosis other than PD by clinical criteria
2. Family history of early onset PD (<age 40) or known personal genetically causal etiology of PD (e.g. SNCA duplication, Parkin, PINK, DJ1) by previously obtained genetic testing
3. Currently pregnant
4. Sarcopenia defined as low BMI (<22 Bahat et al, 2019) with clinically defined weakness
5. Medical history of cardiac arrhythmia, heart failure, stroke / cerebral hemorrhage, epilepsy, other disease of the central nervous system, active cancer, end-stage liver disease, advanced kidney disease (CKD stage 3 or ESRD), beta thalassemia, or any other medical condition deemed by the PI to pose an increased risk for taking part in the study.
6. Inherited or other metabolic disease known to be worsened by ketogenic diet, e.g. inherited defect of lipid or amino acid metabolism
7. Diabetes on SGLT2 inhibitor or uncontrolled diabetes, defined as Hemoglobin A1c > 8.0% on screening test
8. History of kidney stones or gallbladder surgery
9. Biliary / liver disease, defined on screening labs, by presence of any of the following: Total bilirubin (TB) > 2x ULN or > 2 mg/dL; AST >3x ULN; or ALT >5x ULN
10. Uncontrolled hypertension, defined as SBP > 180 mmHg or DBP > 105 mmHg on screening visit
11. Hyperlipidemia defined by LDL >/= 160 mg/dL as per ATP-III guidelines
12. Medical / psychiatric condition identified via clinical assessment in screening visit felt to impede completion of the study*
13. Presence of PD Psychosis or dementia, or other neuropsychiatric or psychiatric illness impeding consent and fidelity to the study intervention and/or measurements
14. Dietary or allergy restrictions as determined by research team to be prohibitive for the study
15. Inability to communicate and provide informed consent in English
16. No history of previous use of ketogenic or similar diet to a degree that could interfere with study blinding

    * A thorough medical and social history will be performed during the screening visit including questions regarding alcohol and substance abuse. If active alcohol abuse or other current substance abuse is identified which could increase the risk of study participation, then participants will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chaudhuri KR, Martinez-Martin P, Brown RG, Sethi K, Stocchi F, Odin P, Ondo W, Abe K, Macphee G, Macmahon D, Barone P, Rabey M, Forbes A, Breen K, Tluk S, Naidu Y, Olanow W, Williams AJ, Thomas S, Rye D, Tsuboi Y, Hand A, Schapira AH. The metric properties of a novel non-motor symptoms scale for Parkinson's disease: Results from an international pilot study. Mov Disord. 2007 Oct 15;22(13):1901-11. doi: 10.1002/mds.21596. PMID 17674410
- [Background] Colla E. Linking the Endoplasmic Reticulum to Parkinson's Disease and Alpha-Synucleinopathy. Front Neurosci. 2019 May 29;13:560. doi: 10.3389/fnins.2019.00560. eCollection 2019. PMID 31191239
- [Background] Chen MJ, Russo-Neustadt AA. Running exercise-induced up-regulation of hippocampal brain-derived neurotrophic factor is CREB-dependent. Hippocampus. 2009 Oct;19(10):962-72. doi: 10.1002/hipo.20579. PMID 19294650
- [Derived] Choi AH, Delgado M, Chen KY, Chung ST, Courville A, Turner SA, Yang S, Airaghi K, Dustin I, McGurrin P, Wu T, Hallett M, Ehrlich DJ. A randomized feasibility trial of medium chain triglyceride-supplemented ketogenic diet in people with Parkinson's disease. BMC Neurol. 2024 Apr 1;24(1):106. doi: 10.1186/s12883-024-03603-5. PMID 38561682
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-N-0153.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited from the pool of participants seen in the NIH Parkinson's Clinic and patients with Parkinson's disease who have participated in other NINDS protocols. Recruitment occurred between January and October 2021.
Pre-assignment Details: Participants were consented and screened for eligibility. 21 participants were screened and 17 participants met eligibility criteria. One participant withdrew after screening but prior to randomization. Eligible participants were randomized in a blinded manner to receive either a Ketogenic diet supplemented with MCT oil or a Standard American Diet x 6 days while an inpatient. This was followed by both groups receiving a Ketogenic Diet supplemented with MCT oil at home x 2 weeks (unblinded).
Groups:
- Ketogenic Diet: Participants consumed a ketogenic diet supplemented with MCT oil x 6 days (inpatient) during phase 1, followed by a 2 week ketogenic diet supplemented with MCT oil (at home) during phase 2.
- Standard American Diet: Participants consumed a standard American diet x 6 days (inpatient) during phase 1, followed by a 2 week ketogenic diet supplemented with MCT oil (at home) during phase 2.
Period: Phase 1 - Inpatient (Blinded)
Arm/Group | Ketogenic Diet | Standard American Diet
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0
Period: Phase 2 - At Home (Unblinded)
Arm/Group | Ketogenic Diet | Standard American Diet
Started | 7 | 9
Completed | 7 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketogenic Diet | Standard American Diet | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibiilty of Ketogenic Diet - Retention (Co-primary Endpoint)
Description: Analysis of feasibility was determined by 3 co-primary endpoints: retention, adherence, and acceptability, measured at the end of week 3 (outpatient segment). After each co-primary endpoint was calculated, three benchmark criteria were used to determine feasibility. All criteria must be met for feasibility to be positive.
  Benchmark criteria for Retention was defined as a completion rate at study end (week 3) of >80%, i.e., >80% of participants must remain in the study at the 3 week time point.
Time Frame: Week 3
Population: Number of participants remaining in the study at week 3.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants consumed a ketogenic diet supplemented with MCT oil (at home) for two weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants | 15

2. Primary Outcome: Feasibility of Ketogenic Diet - Adherence (Co-primary Endpoint)
Description: Analysis of feasibility was determined by 3 co-primary endpoints: retention, adherence, and acceptability, measured at the end of week 3 (outpatient segment). After each co-primary endpoint was calculated, three benchmark criteria were used to determine feasibility. All criteria must be met for feasibility to be positive.
  Benchmark criteria for Adherence was defined as a mean net carbohydrate intake of </=10% during the 2 week outpatient period. Mean net carbohydrate intake was determined using the following calculation: (total carbohydrates minus total dietary fiber) x 4 divided by total calories.
Time Frame: Week 3
Population: Average net carbohydrate intake across all participants during the 2 week outpatient period.
Measure: Mean (Standard Deviation); unit: percentage of diet
Arm/Group | All Participants
Number analyzed (Participants) | 15
percentage of diet | 9.7 (3.2)

3. Primary Outcome: Feasibility of Ketogenic Diet - Acceptability (Co-primary Endpoint)
Description: Analysis of feasibility was determined by 3 co-primary endpoints: retention, adherence, and acceptability, measured at the end of week 3 (outpatient segment). After each co-primary endpoint was calculated, three benchmark criteria were used to determine feasibility. All criteria must be met for feasibility to be positive.
  Acceptability was defined via an exit survey (at end of study week 3) using a 4-point Likert scale to indicate how likely the participant would continue the diet on at least an intermittent basis in the future with 1 representing "Very likely" and 4 representing "Very unlikely". The benchmark criteria for Acceptability was defined as at least 2 out of 4 on the Likert scale.
Time Frame: Week 3
Population: Average score on the Likert scale for diet acceptability across all participants at week 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 15
score on a scale | 2.26 (0.96)

4. Secondary Outcome: Timed Up and Go (TUG)
Description: The Timed Up and Go (TUG) test is a simple test used to assess a person's mobility. The TUG measures the time required to perform a sequence of activities, i.e.,sit-to-stand transfer, straight walking, turning, and walk-to-sit transfer. The TUG is administered at baseline, and each day during the inpatient visit. The results represent a comparison of the group mean score at the end of admission (day 7) for the two cohorts, i.e., patients receiving a Ketogenic Diet and patients receiving a Standard American Diet. A time of greater than 13.5 seconds may suggest a greater risk of falls.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Ketogenic Diet | Standard American Diet
Number analyzed (Participants) | 7 | 9
Seconds | 8.4 (1.2) | 9.1 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected with start dates occurring any time after informed consent was obtained until 7 days (for non-serious AE) or 30 days (for SAEs) after the last day of study participation.
Groups:
- Ketogenic Diet - Phase 1: Participants consumed a ketogenic diet supplemented with MCT oil x 6 days (inpatient) during phase 1.
- Standard American Diet - Phase 1: Participants consumed a standard American diet x 6 days (inpatient) during phase 1.
- Ketogenic Diet - Phase 2: Participants consumed a ketogenic diet supplemented with MCT oil x for 2 weeks (home) during phase 2.
Arm/Group | Ketogenic Diet - Phase 1 | Standard American Diet - Phase 1 | Ketogenic Diet - Phase 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 1/15
Other Adverse Events (participants affected / at risk) | 7/7 | 6/9 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketogenic Diet - Phase 1 (N=7) | Standard American Diet - Phase 1 (N=9) | Ketogenic Diet - Phase 2 (N=15)
Pulmonary Embolus (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketogenic Diet - Phase 1 (N=7) | Standard American Diet - Phase 1 (N=9) | Ketogenic Diet - Phase 2 (N=15)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle ache with headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Indegestion with acid reflux (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Headache s/p hit head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Increased salivation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (increased from baseline) (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flexing and External rotation of toes (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT04584346/Prot_SAP_000.pdf